CLINICAL TRIAL: NCT00370487
Title: Complication Rates of First-Trimester Manual Vacuum Aspiration Abortion Performed by Physicians and Midlevel Providers (MLP) in South Africa and Viet Nam: a Randomised, Controlled, Equivalence Trial.
Brief Title: Comparison of the Safety of First Trimester Abortions Performed by Physicians and Non-Physicians in South Africa and Viet Nam.
Status: Completed | Type: Observational
Sponsor: World Health Organization (Other)
Collaborators: University of Cape Town (Other); Hanoi Obstetrics and Gynecology Hospital (Other)
Other Study IDs: A15324;A15325
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2006-09-06 (Estimated); Status verified 2005-06

CONDITIONS: Abortion, Induced
Keywords: Abortion; Midlevel providers; South Africa; Viet Nam

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
There have been no studies in developing countries assessing the safety of midlevel providers (MLP) compared to physicians in performing first-trimester manual vacuum aspiration abortion. In South Africa and Viet Nam, MLP (midwives and physician assistants) are trained and accredited to perform first trimester abortions to increase women's access to safe abortion services. To assess the safety of abortions performed by midlevel provider compared to physicians, complication rates of first-trimester manual vacuum aspiration are compared between types of providers in the two countries. We test the null hypothesis that the two types of providers provide abortions equally safely.

DETAILED DESCRIPTION:
Objective

There have been no studies in developing countries assessing the safety of midlevel providers (MLP) compared to physicians in performing first-trimester manual vacuum aspiration abortion. In South Africa and Viet Nam, MLP (midwives and physician assistants) are trained and accredited to perform first trimester abortions to increase women's access to safe abortion services. Complication rates of first-trimester manual vacuum aspiration are compared between types of providers in the two countries.

Methods:

A randomized, two-sided controlled equivalence trial was conducted to compare rates of abortion complications. An a priori margin of equivalence of 4.5% with 80% power and a 95% CI ( = 0.025) was used. Women presenting for an induced abortion at up to 12 weeks' gestation were randomly assigned to a physician or a midlevel provider for manual vacuum aspiration and followed-up 10 to 14 days later. Complications were recorded during the abortion procedure, before discharge from the clinic and at follow-up. The study included 25 providers and 2894 cases, 1160 in South Africa and 1734 in Viet Nam.

Results:

Complication rates were 1.4 per 100 for MLP and 0 for physicians in South Africa. In Viet Nam, complication rates were 1.2 per 100 for MLP and 1.1 per 100 for physicians. In both countries, complication rates satisfied the pre-determined statistical criteria for equivalence. In South Africa, the difference in complication rates for mid-level providers and physicians was 1.4 per 100 (CI=0.4 to 2.7). In Viet Nam, the difference in complication rates for mid-level providers and physicians was 0.1 per 100 (CI= -1.0 to 1.2). There were no major immediate complications. Delayed complications were retained products and infection.

Conclusions:

First trimester manual vacuum aspiration abortions performed by trained and accredited midlevel providers in South Africa and Viet Nam were comparable in safety to those performed by physicians. Given appropriate training, midlevel health care providers can provide first trimester manual vacuum aspiration abortions as safely as physician abortion providers.

ELIGIBILITY:
Inclusion Criteria:

* gestation of no more than 12 weeks as estimated by pelvic examination and date of LMP
* age 18 or above
* residence within the catchment area specified for each clinic
* willing to return to clinic for follow-up visit or agree to a telephone or home-based interview
* be able to understand the information given to them and to make personal decisions on whether or not to participate in the study as determined by the study staff
* consent given to participate in the study and consent form signed

Exclusion Criteria:

* uterine sizing of beyond 12 weeks gestation
* under age 18
* unwilling or unable to return to clinic for follow-up visit.
* unwilling to provide consent for participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2860
Dates: Start 2003-09; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hoffman, M.D., Principal Investigator — Women's Health Research Unit, School of Public Health and Family Medicine, Faculty of Health Sciences, University of Cape Town, South Africa; ND Vy, MD, Principal Investigator — National Hospital of Obstetrics and Gynecology, 43 Trang Thi, Hanoi, Viet Nam; My Huong Nguyen, MD, Study Director — National Hospital of Obstetrics and Gynecology, 43 Trang Thi, Hanoi, Viet Nam; Jane Harries, PhD, Study Director — Women's Health Research Unit, School of Public Health and Family Medicine, Faculty of Health Sciences, University of Cape Town, South Africa.